CLINICAL TRIAL: NCT05360524
Title: Laminectomy Alone Versus Laminectomy and Fusion for Traumatic Cervical Spinal Cord Injury Without Instability: A Randomized Controlled Trial
Brief Title: Laminectomy Alone Versus Laminectomy and Fusion for Traumatic Cervical Spinal Cord Injury Without Instability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Sayed Hamed Mohammed, Physician, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Laminectomy vs fusion
Record Dates: First submitted 2022-04-05; First posted 2022-05-04 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Cervical Spinal Cord Injury
MeSH Terms: interventions — Gene Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laminectomy alone in patients with traumatic cervical spinal cord injury without instability (Active Comparator): laminectomy only with expected less operative time, blood loss and restriction of neck motion (compared to laminectomy with fusion). Instrumented fusions also entail the risks of screw misplacement, pseudoarthrosis, distal junction kyphosis, and adjacent segment pathology.
  Interventions: Procedure: Laminectomy alone versus laminectomy and fusion
- Laminectomy and fusion in patients with traumatic cervical spinal cord injury without instability (Active Comparator): Multi-level laminectomy compromises the posterior tension band and increases the mobility of the neck, resulting in post laminectomy kyphosis and potential dynamic injury to the spinal cord . In contrast, spinal instrumentation and fusion helps to eliminate movement at the treated levels and reduce spinal cord tension with less incidence of kyphosis.
  Interventions: Procedure: Laminectomy alone versus laminectomy and fusion

INTERVENTIONS:
Procedure: Laminectomy alone versus laminectomy and fusion — laminectomy only with expected less operative time, blood loss and restriction of neck motion (compared to laminectomy with fusion). Instrumented fusions also entail the risks of screw misplacement, pseudoarthrosis, distal junction kyphosis, and adjacent segment pathology.
  Multi-level laminectomy compromises the posterior tension band and increases the mobility of the neck, resulting in post laminectomy kyphosis and potential dynamic injury to the spinal cord . In contrast, spinal instrumentation and fusion helps to eliminate movement at the treated levels and reduce spinal cord tension with less incidence of kyphosis.

SUMMARY:
The aim of study is to compare clinical and radiological outcomes of laminectomy alone to laminectomy and fusion in the treatment of traumatic cervical spinal cord injury without instability.

DETAILED DESCRIPTION:
Cervical spinal cord injury (CSCI) without instability tends to be caused by a hyperextension force to the neck. This type of injury has been increasing as the elderly population is dramatically increasing.

Although surgery has become the preferred method for management of traumatic unstable cervical spine injury, the treatment of spinal cord injury (SCI) without instability such as fracture, dislocation, and ligamentous injury, however, remains controversial.

Before deciding for surgical or conservative treatment, one should understand the pathophysiology of SCI. Traumatic SCI is dependent on primary damage, such as the dynamic mechanistic force and static pre-existing or concurrent cord compression, and secondary damage, such as edema, ischemia, and inflammation, which lead to demyelination of axons, apoptosis of neural cells, and glial scar formation in the spinal cord.

Advocates of conservative treatment believe that decompression is not effective here, because the compression may have existed before the injury in asymptomatic patients. Therefore, the symptoms develop after a CSCI without instability are probably not a result of the compression itself. On the other hands advocates of surgical treatment believe that decompression could prevent secondary cord damage due to the vicious cycle of "ischemia-edema-ischemia". However, faced with a patient with neurologic dysfunction MRI evidence of cervical spinal cord compression, decompressive surgery is a practical treatment option.

Since these injuries are stable, why to add fusion to laminectomy when it is possible to perform laminectomy only with expected less operative time, blood loss and restriction of neck motion (compared to laminectomy with fusion). Instrumented fusions also entail the risks of screw misplacement, pseudoarthrosis, distal junction kyphosis, and adjacent segment pathology.

Multi-level laminectomy compromises the posterior tension band and increases the mobility of the neck, resulting in post laminectomy kyphosis and potential dynamic injury to the spinal cord . In contrast, spinal instrumentation and fusion helps to eliminate movement at the treated levels and reduce spinal cord tension with less incidence of kyphosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with traumatic cervical spine cord injury admitted to Assiut University Hospital - Department of Orthopaedic and Trauma Surgery regardless of age, mechanism of injury or neurological status changes.

Exclusion Criteria:

1. Associated cervical spine bony or ligamentous injury.
2. Associated primary focal anterior compression of the cervical spinal cord (clear disc herniation).
3. Associated head injury.
4. Kyphotic cervical spine as measured by C2-C7 Cobb angle on X-ray.
5. Previous surgery of the cervical spine.
6. Patients who refuse to participate in the study
7. Patients who are mentally incompetent or unable to comply with the one year follow up regimen

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Neurological recovery. | 3, 6 and 12 month after treatment.
  It is assessed by the improvement (changes) in American Spinal Injury Association (ASIA) motor score). it is based on the motor function score of the 10 pairs of key muscles in the upper and lower limbs, with 5 points for each muscle and 100 points in total.

SECONDARY OUTCOMES:
Neck pain . | 3, 6 and 12 month after treatment.
  It is assessed by the 100 mm visual analog scale (VAS) score (neck).
C2-C7 Cobb angle | 3, 6 and 12 month after treatment.
  C2-C7 Cobb angle< 10°
C7 slope | 3, 6 and 12 month after treatment
  C7 slope <10°, the angle between the horizontal plane and the plane of the superior endplate of the C7 vertebral body.
C2-C7 sagittal vertical axis | 3, 6 and 12 month after treatment
  C2-C7 sagittal vertical axis < 4cm, the anterior offset of C2 from C7.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Mohamed Hassan, Professor, Study Chair — Assiut University
Locations (1):
- Faculty of Medicine Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kawano O, Ueta T, Shiba K, Iwamoto Y. Outcome of decompression surgery for cervical spinal cord injury without bone and disc injury in patients with spinal cord compression: a multicenter prospective study. Spinal Cord. 2010 Jul;48(7):548-53. doi: 10.1038/sc.2009.179. Epub 2010 Jan 12. PMID 20065985
- [Background] Chikuda H, Ohtsu H, Ogata T, Sugita S, Sumitani M, Koyama Y, Matsumoto M, Toyama Y; OSCIS investigators. Optimal treatment for spinal cord injury associated with cervical canal stenosis (OSCIS): a study protocol for a randomized controlled trial comparing early versus delayed surgery. Trials. 2013 Aug 7;14:245. doi: 10.1186/1745-6215-14-245. PMID 23924165
- [Background] McDonald JW, Sadowsky C. Spinal-cord injury. Lancet. 2002 Feb 2;359(9304):417-25. doi: 10.1016/S0140-6736(02)07603-1. PMID 11844532
- [Background] Lee HJ, Kim HS, Nam KH, Han IH, Cho WH, Choi BK. Neurologic Outcome of Laminoplasty for Acute Traumatic Spinal Cord Injury without Instability. Korean J Spine. 2013 Sep;10(3):133-7. doi: 10.14245/kjs.2013.10.3.133. Epub 2013 Sep 30. PMID 24757474
- [Background] Passias PG, Vasquez-Montes D, Poorman GW, Protopsaltis T, Horn SR, Bortz CA, Segreto F, Diebo B, Ames C, Smith J, LaFage V, LaFage R, Klineberg E, Shaffrey C, Bess S, Schwab F; ISSG. Predictive model for distal junctional kyphosis after cervical deformity surgery. Spine J. 2018 Dec;18(12):2187-2194. doi: 10.1016/j.spinee.2018.04.017. Epub 2018 Apr 27. PMID 29709551
- [Background] Fehlings MG, Santaguida C, Tetreault L, Arnold P, Barbagallo G, Defino H, Kale S, Zhou Q, Yoon TS, Kopjar B. Laminectomy and fusion versus laminoplasty for the treatment of degenerative cervical myelopathy: results from the AOSpine North America and International prospective multicenter studies. Spine J. 2017 Jan;17(1):102-108. doi: 10.1016/j.spinee.2016.08.019. Epub 2016 Sep 3. PMID 27597512
- [Background] ASIA and ISCoS International Standards Committee. The 2019 revision of the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI)-What's new? Spinal Cord. 2019 Oct;57(10):815-817. doi: 10.1038/s41393-019-0350-9. Epub 2019 Sep 17. No abstract available. PMID 31530900